CLINICAL TRIAL: NCT02450227
Title: Carotenoid Absorption and Metabolism From Green-leafy Vegetable Matrices - a Explorative Study in Short-bowel Patients and Healthy Controls - The "Popeye-study"
Brief Title: Carotenoid Absorption and Metabolism From Green-leafy Vegetable Matrices
Acronym: Popeye
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is considered non-achievable to recruit the target number of subjects in the short bowel group (n = 12). 10 participants were recruited.
Sponsor: University of Copenhagen (Other)
Collaborators: Agroscope Liebefeld-Posieux Research Station ALP (Other); Rigshospitalet, Denmark (Other); Herta Messerli Stiftung (Unknown); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M220; H-3-2014-112/46407 (Other: The Danish Ethics Committee)
Record Dates: First submitted 2015-05-17; First posted 2015-05-21 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Ileostomy; Functional Disturbance; Healthy
MeSH Terms: interventions — Lutein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinach - Whole leaf (10 mg lutein) (Active Comparator): 1-2: Group given whole leaf as first intervention Whole leaf spinach (10 mg lutein) given every second day for a 15 days period.
  Followed by:
  Minced spinach (10 mg lutein) given every second day for a 15 days period.
  Interventions: Dietary Supplement: Spinach - Whole leaf (10 mg lutein); Dietary Supplement: Spinach - Minced (10 mg/lutein)
- Spinach - Minced (10 mg lutein) (Experimental): 2-1: Group given minced spinach as first intervention Minced spinach (10 mg lutein) given every second day for a 15 days period.
  Followed by:
  Whole leaf spinach (10 mg lutein) given every second day for a 15 days period.
  Interventions: Dietary Supplement: Spinach - Whole leaf (10 mg lutein); Dietary Supplement: Spinach - Minced (10 mg/lutein)

INTERVENTIONS:
Dietary Supplement: Spinach - Whole leaf (10 mg lutein) — Identical spinach meals processed in two different ways by Frigodan, served alone or together with habitual diet
Dietary Supplement: Spinach - Minced (10 mg/lutein) — Identical spinach meals processed in two different ways by Frigodan, served alone or together with habitual diet

SUMMARY:
Absorption and metabolism of carotenoids from two types of spinach preparations will be investigated in two study groups, short bowel/ileostomy and healthy, respectively.

The study will be conducted as a randomised, controlled, 2-way crossover study in 24 participants (12 in each group), randomized to two sequences (1-2, 2-1) of interventions with a more and a less bio-accessible spinach preparation. The serum, chylomicron and fecal/effluent levels of lutein and beta-carotene will be determined.

DETAILED DESCRIPTION:
Absorption and metabolism of carotenoids from two types of spinach preparations will be investigated in two study groups, short bowel/ileostomy and healthy, respectively.

The study will be conducted as a randomised, controlled, 2-way crossover study. Twenty four participants (12 in each group) will be randomized to two sequences (1-2, 2-1) of interventions with a more and a less bio-accessible spinach preparation (differentiates only on the basis of particle size).

The intervention period is sub-divided into three parts: run-in period (48 hours) with a standardized low-carotenoid diet, 0-24 hours (follow-up period 1 (FP1)) and 24 hours - 2 weeks (FP2). The intervention periods will be separated by a wash-out period of at least 14 days.

At start of each intervention, the intervention meal (breakfast) is served, followed by standardized, carotenoid-free meals in the following 24 hours. Participants will in FP1 and FP2 receive an intervention meal every second day. Participants will otherwise keep their habitual diets during these follow-up periods.

Study participants are asked to collect urine during 24 hours before and after the first intervention meal in each period. They will also collect feces/ileostomy efflux for 24 hours before and after initiation of the intervention for short bowel/ileostomy patients and for 48 periods in the healthy volunteers, respectively. Overnight-fasting serum samples are drawn at day 1, 7 and 15 of each intervention period. On day 1 plasma samples are drawn at 0,1, 3, 4, 6, 7, 9 and 24 hours post first intervention meal.

Plasma and effluent levels of lutein and beta-carotene will be determined and chylomicrons are also separated from these samples for determination of carotenoids.

Volunteers also have their macula examined for density of the yellow spot before and after the intervention. Plasma and effluent levels of other carotenoids as well as fat-soluble vitamins are also determined. The samples will also be subjected to metabolic profiling for further exploration and hypothesis generation.

ELIGIBILITY:
List of inclusion criteria:

* Healthy adults (18-80 years old)
* Body Mass Index (BMI) between 18,9-28
* Normal fasting blood glucose (BS) (1,9-5,6 mmol/L)
* Tolerates: Potatoes, rice, chicken, meat (non vegan/vegetarian).

List of exclusion criteria:

* Intestinal diseases (among healthy controls), systemic infections, psychiatric disorders, metabolic diseases (incl. diabetes), and any clinical condition/circumstance which assessed by the study official makes the person unfit for participation in the trial.
* Patients diagnosed with short bowel syndrome (SBS).
* Chronic or frequent use of medication. Primarily consumption of drugs with known effect/side effects on fat absorption. Further, anticoagulants (Marevan) and systemic treatment with glucocorticoids.
* Have or have had a drug addiction
* Smokers
* Alcohol consumption beyond the recommended (7/14 units per week for women/men, respectively)
* Intake of vitamins or other supplements (3 months before the study and during the study) (healthy controls). Subjects from the patient group included only with stable intake of dietary supplements through the last 3 months.
* Sampling or donation of larger amount of blood e.g. as blood donors or to other scientific experiments from 3 months before the study until its completion.
* allergy or intolerance to any of the foods included in the study.
* Women who are nursing, pregnant or planning pregnancy
* Not able to comply with the procedures protocol.
* Macular degeneration to a degree greeter than or equal to a surface area with one or more drusen larger than 125 microns in diameter in at least one eye.
* Cataracts, macular- or other ocular disease, preventing depiction of xanthophyll pigment.

The following separate registered information was additionally recorded for short bowel/ileostomy patients:

* Time since operation (stable, >1 year post operation)
* Type of disease/background for operation
* Intestinal anatomy (inclusive length and type of residual intestine)
* Type and doses of vitamin and other types of supplementation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum concentration of lutein and beta-carotene | 15 days
  Difference in serum concentration of lutein and beta-carotene between baseline and the end of each intervention period.

SECONDARY OUTCOMES:
Concentration of lutein and beta-carotene in the chylomicron/TLR fraction | 24 hours
  Changes in concentration of lutein and beta-carotene in the chylomicron/TLR fraction (area under the curve, AUC) 24 hours post first intervention meal in each intervention periods.
Total lutein and beta-carotene sekretion with feces/ileostomy-efflux | 48/24 hours
  Total lutein and beta-carotene sekretion with feces/ileostomy-efflux 48 and 24 hours postprandial, for healthy and ileostomy patients, respectively.
Concentration of other carotenoids in the chylomicron/TLR fraction | 24 hours
  Changes in concentration of other carotenoids in the chylomicron/TLR fraction (area under the curve, AUC) 24 hours post first intervention meal in each intervention periods.
Serum concentration of other carotenoids | 15 days
  Difference in serum concentration of other carotenoids between baseline and the end of each intervention period.
Serum concentration of other fat-soluble vitamins | 15 days
  Difference in serum concentration of other vitamins (A, E; D, K) between baseline and the end of each intervention period.
Changes in metabolic markers | 24 hours
  Changes in overall metabolic markers from urine 24 hours postprandial
Changes in metabolic markers | 24 hours
  Changes in overall metabolic markers in the chylomicron/TLR fraction 24 hours postprandial
Changes in metabolic markers | 15 days
  Changes in overall metabolic markers in serum at the end of each intervention period.
Level of optical density of the macula lutea | Baseline
  Level of optical density in the macula lutea (MPOD), in the spectra where xanthophyll pigment is absorbing light.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Rigshospitalet, Department of Gastroenterology, CA-2121, Copenhagen Ø
  - Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg C